CLINICAL TRIAL: NCT06384976
Title: KYSA-7: A Phase 2, Open-Label, Randomized, Multicenter Study of KYV-101, an Autologous Fully Human Anti-CD19 Chimeric Antigen Receptor T-Cell (CD19 CAR T) Therapy, in Subjects With Refractory Primary and Secondary Progressive Multiple Sclerosis
Brief Title: KYSA-7: A Study of Anti-CD19 CAR T-Cell Therapy, in Subjects With Refractory Primary and Secondary Progressive Multiple Sclerosis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kyverna Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KYSA-7; KYV101-007 (Other: Kyverna Therapeutics)
Record Dates: First submitted 2023-11-21; First posted 2024-04-25 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Multiple Sclerosis, Primary Progressive; Multiple Sclerosis, Secondary Progressive; Multiple Sclerosis; MS
Keywords: KYV-101; multiple sclerosis; autoimmune disease; anti-CD19 CAR-T therapy; cellular therapy; MS
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive; Multiple Sclerosis; Autoimmune Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- KYV-101 CAR-T cells with lymphodepletion conditioning (Experimental): Dosing with KYV-101 CAR T cells
  Interventions: Biological: KYV-101; Drug: Standard lymphodepletion regimen
- Anti- CD20 mAb (Active Comparator): Dosing with anti-CD20 mAb
  Interventions: Drug: Anti-CD20 mAB

INTERVENTIONS:
Biological: KYV-101 — Anti-CD19 CAR-T cell therapy
  Arms: KYV-101 CAR-T cells with lymphodepletion conditioning
Drug: Standard lymphodepletion regimen — CYC/FLU
  Arms: KYV-101 CAR-T cells with lymphodepletion conditioning
Drug: Anti-CD20 mAB — Anti-CD20 mAB
  Arms: Anti- CD20 mAb

SUMMARY:
A Study of Anti-CD19 Chimeric Antigen Receptor T-Cell (CD19 CAR T) Therapy, in Subjects with Refractory Primary and Secondary Progressive Multiple Sclerosis

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is an autoimmune and neurodegenerative disease in which lymphocytes at first attack the myelin sheaths within the central nervous system (CNS), accompanied or later followed by axonal damage. B cells play a central and multifunctional role in the immunopathogenesis of MS. B cells present antigen to T cells in stimulating a pro-inflammatory immune cascade, secrete pathogenic cytokines, moderate T cell and myeloid cell functions, form structural B cell meningeal follicles within the human central nervous system and produce pathogenic antibodies upon evolution to plasma cells.

CD19-targeted chimeric antigen receptor (CAR) T cells harness the ability of cytotoxic T cells to directly and specifically lyse target cells to effectively deplete B cells in the circulation and in lymphoid and potentially non-lymphoid tissues. KYV-101, a fully human anti-CD19 CAR T-cell therapy, will be investigated in adult subjects with refractory primary and secondary progressive multiple sclerosis.

ELIGIBILITY:
Key Inclusion Criteria:

1. Subject must have a history of diagnosis of primary progressive or secondary progressive MS.
2. History of treatment with anti-CD20 mAb with continuing evidence of worsening physical disability over a period of ≥6 months, with documented clinical disability progression within the 2 years prior to inclusion.

Key Exclusion Criteria:

1. Monophasic disease, radiologically isolated syndrome, clinically isolated syndrome, progressive solitary sclerosis or relapsing-remitting disease as defined by the 2017 McDonald criteria.
2. History of CNS or spinal cord tumor, metabolic or infectious cause of myelopathy, genetically inherited progressive CNS disorder, sarcoidosis, non-MS progressive neurologic condition or PML.
3. Prior treatment with cellular therapy (CAR-T) or gene therapy product directed at any target
4. History of allogeneic or autologous stem cell transplant
5. Evidence of active hepatitis B or hepatitis C infection
6. Positive serology for HIV
7. Primary immunodeficiency
8. History of splenectomy
9. History of stroke, seizure, dementia, Parkinson's disease, coordination movement disorder, cerebellar diseases, psychosis, paresis, aphasia, and any other neurologic disorder investigator considers would increase the risk for the subject
10. Impaired cardiac function or clinically significant cardiac disease
11. Previous or concurrent malignancy with the following exceptions:

    1. Adequately treated basal cell or squamous cell carcinoma (adequate wound healing is required prior to screening)
    2. In situ carcinoma of the cervix or breast, treated curatively and without evidence of recurrence for at least 3 years prior to screening
    3. A primary malignancy which has been completely resected, or treated, and is in complete remission for at least 5 years prior to screening

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-09-20 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate efficacy of KYV-101 | at least 12 weeks
  Confirmed disability Progression on the EDSS scale. The EDSS scale ranges from 0 to 10 in 0.5- unit increments that represent higher levels of disability. Scoring is based on an examination by a neurologist.

SECONDARY OUTCOMES:
To characterize the safety and tolerability of KYV-101 | Up to 2 years
  Incidence and severity of adverse events (AEs)
To characterize the safety and tolerability of KYV-101 | Up to 2 years
  Incidence and severity of adverse events of special interests (AESIs)
To characterize the safety and tolerability of KYV-101 | Up to 2 years
  Incidence and severity of serious adverse events (SAEs)
To evaluate efficacy of KYV-101 | up to 12 weeks
  Composite Confirmed Disability Progression (CCPD)
To characterize the pharmacokinetics (PK) | Up to 2 years
  Levels of Chimeric antigen receptor positive (CAR-positive) T cell counts
To characterize the pharmacokinetics (PK) | Up to 2 years
  Levels of CAR Transgene levels
To characterize the Pharmacodynamics (PD) | Up to 2 years
  Levels of B cell in the blood
To characterize the Pharmacodynamics (PD) | Up to 2 years
  Serum cytokines will be measured by multiplexed mesoscale discovery (MSD) assay and will include cytokines historically associated with potential CAR T toxicity (CRS and ICANS) such as gamma interferon (IFNg) and interleukin 6 (IL-6).
To evaluate the immunogenicity (humoral response) of KYV-101 | Up to 2 years
  Percentage of participants who develop anti-KYV-101 antibodies by immunoassays)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Kyverna Therapeutics, Inc.
Locations (1):
- Stanford University Medical Center, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Silva BA, Miglietta E, Ferrari CC. Insights into the role of B cells in the cortical pathology of Multiple sclerosis: evidence from animal models and patients. Mult Scler Relat Disord. 2021 May;50:102845. doi: 10.1016/j.msard.2021.102845. Epub 2021 Feb 16. PMID 33636613